CLINICAL TRIAL: NCT04836611
Title: Cannabinoides Concentrations and Hyperemesis Syndrom Occurrence in Regular Cannabis Consumer (CANEMESE)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Poitiers University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: CANEMESE
Record Dates: First submitted 2021-03-29; First posted 2021-04-08 (Actual); Last update posted 2021-10-06 (Actual); Status verified 2021-09

CONDITIONS: Chronic Consumption of Cannabis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- regular cannabis consumer patients (Other)
  Interventions: Procedure: 1 blood sample

INTERVENTIONS:
Procedure: 1 blood sample — 2 groups of subjects (group 1 : with diagnosis of CHS - group 2 : no diagnosis of CHS) will have 2 blood and 1 urine samples + 1 questionnaire
  Other Names: 1 urine sample

SUMMARY:
The Cannabinoide Hyperemesis Syndrom (CHS) is defined as a recurrent syndrome of intractable vomiting that occurs in chronic cannabis consumers. The diagnosis is linked to clinical criteria only. The physiopathology of CHS is unknown and we observe an increase of cases with this syndrom since 2016 (Schreck et al., 2018).

The aim of this study is to investigate the involvement of exogenous cannabinoids concentrations in chronic cannabis users in the occurrence of CHS.

ELIGIBILITY:
Inclusion Criteria:

* Subjects without protection by a legal regime (guardianship, trusteeship)
* Subjects affiliated to an appropriate social security system
* Subjects must sign an informed consent form

Inclusion Criteria for Group 1:

- Subjects must have the CHS diagnosis confirmed

Inclusion Criteria for Group 2:

- Subjects must be chronic cannabis consumers and never had CHS

Exclusion Criteria:

* Subjects must not have addictive comorbidities or psychoactive substance abuse (except alcohol and tabacco)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2021-07-01 (Actual); Primary Completion 2023-06-30 (Estimated); Study Completion 2023-06-30 (Estimated)

PRIMARY OUTCOMES:
involvement of exogenous cannabinoids concentrations in chronic cannabis users in the occurrence of CHS (see details below for exogenous cannabinoids) | on the day of subjects inclusion
  blood and urine concentration, unit of measure ng/mL
THC (Tetrahydrocannabinol) | on the day of subjects inclusion
  blood and urine concentration, unit of measure ng/mL
metabolite of THC : THC-OH (11-hydroxy-Δ⁹-tétrahydrocannabinol) | on the day of subjects inclusion
  blood and urine concentration, unit of measure ng/mL
metabolite of THC : THC-COOH (11-nor-9-carboxy-Δ⁹-tétrahydrocannabinol) | on the day of subjects inclusion
  blood and urine concentration, unit of measure ng/mL
CBD (Cannabidiol) | on the day of subjects inclusion
  blood and urine concentration, unit of measure ng/mL
CBN (Cannabinol) | on the day of subjects inclusion
  blood and urine concentration, unit of measure ng/mL
CBG (Cannabigerol) | on the day of subjects inclusion
  blood and urine concentration, unit of measure ng/mL

CONTACTS AND LOCATIONS:
Locations (1):
- CHU, Poitiers, France

IPD SHARING:
Plan to Share IPD: Undecided